CLINICAL TRIAL: NCT07120607
Title: Clinical Study on the Safety and Efficacy of CD7 CAR-γδT Cell Injection for the Treatment of Relapsed/Refractory Leukemia
Brief Title: Allogeneic CD7 CAR γδ T Cells Therapy Recurrent/Refractory Leukemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xiaoyu Zhu, Director of Hematology Department, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH10601-TAL-01（0）
Record Dates: First submitted 2025-08-05; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Leukemia
Keywords: CAR γδ T cells; CD7 positive; Recurrent refractory
MeSH Terms: conditions — Leukemia | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with relapsed/refractory acute T-cell leukemia/lymphoma and acute myeloid leukemia (Experimental)
  Interventions: Biological: CD7 CAR-γδT cell（QH106）; Drug: Fludarabine (FLU); Drug: Cyclophosphamide (CTX)

INTERVENTIONS:
Biological: CD7 CAR-γδT cell（QH106） — Allogenic CD7 CAR-γδT cell，Intravenous on day0; dose escalation (3+3) : dose 1 (1 × 10^8 CAR+ cells) , dose 2 (3 × 10^8CAR+ cells/kg，dose 3 (6× 10^8 CAR+ cells）;
Drug: Fludarabine (FLU) — Intravenous fludarabine 30~50 mg/m^2/day on days-5, -4, and -3；
Drug: Cyclophosphamide (CTX) — Intravenous cyclophosphamide 500~1000 mg/m^2/day on days -5, -4, and -3.

SUMMARY:
CD7 is highly expressed in T-cell acute lymphoblastic leukemia (T-ALL) and T-cell lymphoma. Approximately 10-30% of cute myeloid leukemia(AML) patients exhibit CD7 expression, particularly in early myeloid progenitor cell-derived AML (e.g., M0/M1 subtypes), mixed-phenotype acute leukemia (MPAL), and AML with high-risk genetic abnormalities (such as TP53 mutations or complex karyotypes). CD7-positive AML patients typically have poor prognosis, poor response to standard chemotherapy, and shorter overall survival (OS). Targeted CD7 cell therapies may represent a promising direction for the treatment of these diseases.

DETAILED DESCRIPTION:
This study is a single-arm,open-label, dose-escalation clinical trial. It is planned to enroll 9-18 patients with CD7-positive relapsed/refractory T-ALL/LBL and relapsed/refractory AML. The study will use a 3+3 design for dose escalation, with three initial dose groups: 1*10^8 CAR+ cells, 3*10^8 CAR+ cells, and 6*10^8 CAR+ cells.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 14 years, no gender restrictions;
2. Diagnosed with TALL/LBL according to the NCCN Acute Lymphoblastic Leukemia Clinical Practice Guidelines (2023.V2); or diagnosed with AML according to the NCCN Acute Myeloid Leukemia Clinical Practice Guidelines (2023.V6);
3. Meet the criteria for relapsed or refractory T-ALL/LBL, including any of the following:

   1. Relapsed: after achieving complete remission(CR), peripheral blood or bone marrow shows >5% blast cells or extramedullary lesions in any site;
   2. Refractory: primary refractory cases that did not achieve CR after standard induction chemotherapy.

   Or meets the criteria for relapsed or refractory AML, including any of the following:
   1. Relapsed: leukemic cells reappear in peripheral blood or ≥5% of blast cells in bone marrow (excluding other causes such as bone marrow regeneration after consolidation chemotherapy) or extramedullary leukemic cell infiltration after achieving CR;
   2. Refractory: primary cases that remain unresponsive after two cycles of standard treatment; Patients who relapse within 12 months after consolidation therapy following CR; patients who relapse after 12 months and are unresponsive to conventional chemotherapy; patients with two or more relapses; patients with persistent extramedullary leukemia;
4. Cytological confirmation of tumor cell immunophenotyping as CD7-positive during screening;
5. Expected survival time exceeding 3 months;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
7. Organ function meets the following requirements:

   * Liver function: ALT ≤ 3 × ULN; AST ≤ 3 × ULN; Total bilirubin ≤ 3.0 × ULN.
   * Renal function must meet the following criteria: serum creatinine ≤ 1.5 × upper limit of normal (ULN);
   * Cardiac function: echocardiogram showing left ventricular ejection fraction ≥ 50%;
   * Pulmonary function: normal oxygen saturation without oxygen supplementation.
8. Female participants of childbearing potential and male participants whose partners are of childbearing potential must use medically approved contraceptive measures or abstain from sexual intercourse during the study treatment period and for at least 6 months after the study treatment period. Female participants of childbearing potential must have a negative serum HCG test within 7 days prior to study enrollment and must not be breastfeeding.
9. No significant genetic disorders;
10. The subject or their legal guardian voluntarily participates in this study, understands the trial information, objectives, and risks described in the informed consent form, and can provide a signed and dated informed consent form;
11. The subject or their legal guardian is willing and able to comply with all trial requirements.

Exclusion criteria:

1. Patients with a history of severe central nervous system disorders, such as uncontrolled epileptic seizures, stroke, severe brain injury with aphasia, paralysis, dementia, Parkinson's disease, or mental disorders;
2. Heart failure classified as NYHA functional class III or IV;
3. Any of the following unstable cardiovascular conditions occurring within the past 6 months prior to screening (including but not limited to): unstable angina, cerebral ischemia or cerebrovascular accident, myocardial infarction, severe arrhythmias requiring medication (such as rapid atrial fibrillation, high-degree atrioventricular block, ventricular tachycardia, ventricular fibrillation, or torsades de pointes); Undergone coronary angioplasty, coronary artery stent implantation, or coronary artery bypass surgery; experienced thrombosis or embolism events (e.g., cerebrovascular events [including transient ischemic attacks, but excluding lacunar cerebral infarction], deep vein thrombosis [excluding deep vein thrombosis caused by PICC catheter placement], pulmonary embolism, etc.);
4. Presence of disseminated intravascular coagulation;
5. Presence of severe autoimmune diseases or immunodeficiency disorders;
6. Presence of active graft-versus-host disease requiring ongoing systemic treatment;
7. Subjects currently receiving systemic steroid or other immunosuppressive therapy prior to screening, and who, as determined by the investigator, will require long-term use of such therapy after enrollment (excluding inhaled or topical use);
8. Other severe medical conditions deemed inappropriate for enrollment by the investigator (e.g., uncontrolled hypertension or diabetes, severe renal insufficiency, severe pulmonary dysfunction, etc.);
9. Active HBV or HCV infection (HBV-DNA positive or HCV-RNA positive), HIV-positive status, or positive syphilis test results;
10. Other severe or persistent active infections;
11. Adverse events related to systemic immunotherapy (including other investigational drugs or medical device interventions) prior to screening have not yet decreased to Grade 1 severity or returned to baseline status;
12. Immunosuppressive agents have been discontinued for less than 2 weeks;
13. Those who have received CAR-T cell therapy in the past;
14. History of allergy to any component of the cell product;
15. Vaccination or any surgical procedure within 4 weeks prior to screening;
16. Other conditions deemed by the investigator to potentially increase the risk to the subject or interfere with trial results.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | 12 months
  AE is defined as any adverse medical event from the date of lymphocyte depletion chemotherapy to 12 months after QH106 infusion. Among them, cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria, graft-versus-host disease (GVHD) according to criteria defined by the Mount Sinai Acute GVHD International Consortium. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0.
Incidence of Dose-Limiting Toxicities (DLTs) | First infusion date of QH106 up to 28 days

SECONDARY OUTCOMES:
Pharmacodynamics: Peak level of cytokines in serum | Up to 28 days after infusion
Pharmacokinetics: Persistence of QH106 | 12 months
  Persistence of QH106 assessed by number in peripheral blood
Overall Response rate (ORR) | 12 months
  CR (complete remission) /CRh (CR with partial hematological recovery) The proportion of subjects who achieved remission /CRi (complete remission with incomplete hematological recovery) /PR (partial remission)
Negative remission rate of minimal residual disease (MRD) in leukemia | 12 month
Duration of remission (DOR) | 12 month
Leukemia-free survival period(LFS) | 12 month
Overall survival (OS) | 12 month
Immunogenicity: Proportion of subjects with anti drug antibody (ADA) | 12 month